CLINICAL TRIAL: NCT03327298
Title: Direct Pedicle Visualization And Disc Space Orientation As The Only Guide For Lumbar Pedicular Screw Insertion
Brief Title: Free Hand Lumbar Pedicular Screw Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hosni Salama, Assistant professor, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#3925-24-3-2014
Record Dates: First submitted 2017-10-17; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Lumbar Spondylolisthesis
Keywords: Pedicle screw. Free hand. Lumbar fixation
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- accuracy of pedicle screw insertion (Other): postoperative CT lumbar spine axial and sagittal views.
  Interventions: Procedure: pedicle screw fixation

INTERVENTIONS:
Procedure: pedicle screw fixation — One hundred forty four screws were placed in the lumbosacral pedicles of 32 patients using free hand technique depending on direct visualization of the pedicles, roots, and intervertebral disc ( IVD) after doing full laminectomy, then postoperative CT was done for evaluation of pedicle violation.

SUMMARY:
Background: Different methods for lumbar pedicular screw insertion have been advocated, however each technique has its cons and pros. Due to limited resources for O-Arm and navigation in our locality, the investigator was enforced to use the surgical skills to minimize the need for such advanced modalities.

Aim of the study: Is to clarify the benefits of the use of free hand technique using direct visualization of the pedicles and disc space as the only guide for pedicular screw insertion using postoperative CT for evaluation of the accuracy of pedicle screw insertion.

Patients and methods: One hundred and forty four screws were inserted in 32 patients using direct pedicle visualization and disc space orientation as a single intraoperative reference guide. The study was conducted in Zagazig University Hospitals from May, 2014 to June, 2015. CT was done for all patients as a direct postoperative evaluation tool.

DETAILED DESCRIPTION:
Patients and methods: This study was conducted in Zagazig University Hospitals in the period from May 2014 to June 2015 after approval from the Zagazig University Institutional Review Board (Zu-IRB). All patients were subjected to complete history talking, clinical evaluation and adequate radiological and laboratory investigations.

The radiological studies included plain X-Ray lumbosacral spine, anteroposterior, lateral neutral, and lateral dynamic views (lateral with flexion and lateral with extension), MRI lumbosacral spine sagittal and axial views, and in some cases CT lumbosacral spine with sagittal reconstruction. All these modalities give us a good idea about both soft tissue and bony pathology in the area of interest. Selection of the patients for surgery was based on clinicoradiologic items.

All the cases of pedicular screw insertion were preceded by full laminectomy with discectomy for interbody fusion. In all cases the medial and inferior aspects of the pedicle are clearly visualized, so selection of the entry point and direct observation of medial and inferior pedicle violation are two main advantages of this technique. On the other hand after discectomy the disc space with the two parallel endplates are available for use as a guide for screw craniocaudal angulation.

After the removal of the whole lamina with its inferior articular processes and removal of fibrocartilagenous tissues overlying the exiting roots and removal of the intervertebral disc, the anatomy of the pedicle and its relation to the exiting roots is clearly evident.

Starting pedicular screw insertion, part of the cortical bone at the inferolateral edge of the superior facet is removed. This entry point lies exactly along the transverse plane passing through the middle of the corresponding transverse process.

At the same time the inferior and medial surfaces of the pedicle along with the exiting nerve root are clearly visualized, so all factors needed for correct pedicle screw insertion are available including the correct entry point, the mediolateral and craniocaudal orientation in addition to the visual protection provided from inside the canal to observe any medial or inferior pedicle violation.

The investigator used to insert a dissector inside the disc space as an additional guide to craniocaudal orientation of the screw which should be parallel to the disc space.

The process of pedicular screw insertion is completed as usual and the disc space is properly curetted using the suitable shavers then the prepared autologous bone graft is impacted in the disc space. The remaining screws are inserted and the rods are installed and secured as usual.

The time needed for each screw insertion was calculated. During the previous steps neither fluoroscopic guidance nor neuronavigation were used.

After completion of the previous steps, a single lateral and anteroposterior film was used to confirm the correct screw position.

The surgery is completed as usual and the patient is discharged for follow up after two weeks, during which a complementary CT scan lumbar spine is routinely performed and analyzed for the accuracy of the screw position.

Pedicle violation was assessed whether medial, inferior, lateral or superior.

ELIGIBILITY:
Inclusion Criteria:

* single level or double level degenerative spondylolisthesis

Exclusion Criteria:

* other causes of spondylolisthesis

Ages: 24 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05-10 (Actual); Primary Completion 2015-06-05 (Actual); Study Completion 2015-06-05 (Actual)

PRIMARY OUTCOMES:
pedicle screw accuracy | 2 weeks
  Pedicle violation was assessed whether medial, inferior, lateral or superior using postoperative CT

IPD SHARING:
Plan to Share IPD: No